CLINICAL TRIAL: NCT04708522
Title: Remote Delivery of a Brief Self-guided Breath Control and Mindfulness Exercise for the Treatment of Post-concussion Anxiety and Depression Symptoms: The Feasibility of a Randomized Control Trial
Brief Title: Breath Control and Mindfulness for Post Concussion Anxiety and Depression: a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 118148
Record Dates: First submitted 2020-12-16; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-11

CONDITIONS: Post-Concussion Syndrome; Anxiety Disorders and Symptoms; Depressive Symptoms
Keywords: Breath control; Mindfulness
MeSH Terms: conditions — Post-Concussion Syndrome; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breath Control (Experimental): Participants in the breath control study arm will be given a breathing exercise that is to be completed in a comfortable upright seated posture. This intervention exercise will be completed daily for a period of 8 weeks.
  Interventions: Behavioral: Breath Control - Equal Breathing Technique
- Guided Mindfulness (Experimental): Participants in the guided mindfulness study arm will be lead through a seated mindfulness exercise. This intervention exercise will be completed daily for a period of 8 weeks.
  Interventions: Behavioral: Guided Mindfulness Exercise
- Control (Sham Comparator): Participants in the control group will receive a sham intervention. The sham intervention will involve minimal instructed meditation exercise. This intervention exercise will be completed daily for a period of 8 weeks.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Breath Control - Equal Breathing Technique — The equal breathing (EB) exercise also known as square or box breathing will follow the four-part breathing cycle of inhalation, hold, exhalation, hold, repeat. Each part of the cycle will be a 4 second count repeated for 20 minutes.
  Arms: Breath Control
Behavioral: Guided Mindfulness Exercise — The guided seated mindfulness (GSM) exercise will lead the participant through a 20 minute mindfulness meditation exercise using an audio recording.
  Arms: Guided Mindfulness
Behavioral: Control — The control intervention will utilize a sham exercise. The participant will be asked to rest in a comfortable seated position for the duration of the 20 minute session.
  Arms: Control

SUMMARY:
Persistent-post-concussion symptoms (PPCS) is a condition that effects on average one in seven persons following a concussion. Anxiety and depression symptoms are experienced by over one-third of those with PPCS. These symptoms can delay recovery from a concussion. Two techniques used to treat anxiety and depression symptoms are breath control and mindfulness exercises. This 8-week feasibility study will evaluate the implementation and compliance of a remote delivered breathing and mindfulness treatment program for individuals experiencing PPCS anxiety or depression symptoms.

DETAILED DESCRIPTION:
This study will assess the feasibility of a randomized control study designed to remotely deliver a breath control and guided mindfulness exercise to individuals experiencing post-concussion symptoms of anxiety or depression. Participants will be randomized into one of the study arms after they have met eligibility criteria and have given informed consent. Study arm interventions include a 20-minute paced breathing (breath control) exercise, a 20-minute guided mindfulness exercise, and a sham control arm that incorporates a minimal instruction 20-minute quiet sitting meditation exercise. The participant is asked to complete their assigned intervention daily for a period of eight weeks and to complete weekly and biweekly follow-up questionnaires. The questionnaires will include the Rivermead Post-Concussion Syndrome Questionnaire (RPQ) and the Positive Affect Negative Affect Survey Short Form (PANAS) completed weekly, the General Anxiety and Depression questionnaire (GAD-7) and the Patient Health Questionnaire (PHQ-9) completed biweekly. These questionnaires will be completed prior to a participant commencing the study (pre-test measure), at weekly intervals throughout the study (at end of week), and at the conclusion of the 8-week study (post-test measure). At the conclusion of the study participants will be asked to complete the Treatment Acceptability / Adherence Scale (TAAS), a measure used to assess the acceptability of the intervention from the point of view of the participant. All participant outcome measures, and intervention tracking questionnaires will be administered through a secure internet user-input interface.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥18 to ≤65 years of age
* Males and females
* Ability to comprehend English (written and spoken)
* Physician-diagnosed concussion ≥ 4weeks prior to commencing study
* Experiencing post-concussion symptoms (>0 on the RPQ)
* Experiencing symptoms of anxiety and/or depression (Score ≥ 5 on the GAD-7 or ≥ 5 on the PHQ-9)
* Access to an internet accessible device (e.g., computer, smart phone or tablet)
* Access to a smart device (iOS or Android) (required for use of "Awesome Breathing" application)

Exclusion Criteria:

* <18 or >65 years of age
* Score < 5 on the GAD-7 or < 5 on the PHQ-9
* Score 0 on RPQ
* Inability to comprehend English (written and/or spoken)
* History of cardiovascular or cardiorespiratory condition
* History of non-traumatic acquired brain injury
* History of neurological or neurodevelopment disorder
* History of unmanaged or managed psychiatric diagnosis (i.e., mental health issue, including bipolar, schizophrenia, etc.)
* No history substance abuse (drug or alcohol)
* Current pregnancy
* Currently attending other yogic or meditation/mindfulness therapy sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Start of recruitment and end of recruitment (approximately 4 months from initiation of study)
  Proportion of screened individuals choosing to participate (and reasons for not participating)
Feasibility of completion | Start of study participation at baseline and end of study participation at completion of study (approximately 6 months from initiation of study)
  Proportion of participants who drop-out prior to program completion
Feasibility of compliance | Start of study participation at baseline and end of study participation at completion of study (approximately 6 months from initiation of study)
  Proportion of program sessions attended (and reasons for non-attendance); proportion of participants that complete surveys
Feasibility of delivery | Start of recruitment and end of study (approximately 6 months from initiation of study)
  Investigator time-cost analysis of intervention delivery (investigator time/participant)
Acceptability of intervention | Assessed at conclusion of 8-week intervention participation for duration of study
  Evaluated using Treatment Acceptability/Adherence Scale - individual item mean score of 10 item questionnaire each ranging from 1 (strongly disagree) to 7 (agree strongly)
Effectiveness of intervention (PHQ-9) | Assessed at baseline, at the end of weeks 2, 4, 6, and 8 throughout intervention participation for duration of study
  Change in participant outcome measures (questionnaires) for all treatment arms:
  Change in depressive symptoms measured by PHQ-9 - total score ranges from 0 (no symptoms) to 27 (severe symptoms) for all treatment arms
Effectiveness of intervention (GAD-7) | Assessed at baseline, at the end of weeks 2, 4, 6, and 8 throughout intervention participation for duration of study
  Change in participant outcome measures (questionnaires) for all treatment arms:
  Change in anxiety symptoms measured by GAD-7 - total score ranges from 0 (no symptoms) to 21 (severe symptoms) for all treatment arms
Effectiveness of intervention (RPQ) | Assessed at baseline, at the end of weeks 1, 2, 3, 4, 5, 6, 7 and 8 throughout intervention participation
  Change in participant outcome measures (questionnaires) for all treatment arms:
  Change in post-concussion symptoms measured by RPQ - total score ranges from 0 (not experienced) to 64 (severe problem) for all treatment arms
Effectiveness of intervention (PANAS) | Assessed at baseline, at the end of weeks 1, 2, 3, 4, 5, 6, 7 and 8 throughout intervention participation
  Change in participant outcome measures (questionnaires) for all treatment arms:
  Change in positive and negative affect measured by PANAS - total score ranges from 10 (lower) to 50 (higher) for each of positive affect and negative affect for all treatment arms

SECONDARY OUTCOMES:
Participant demographic data | Baseline
  Participant demographic data will be used to describe participant volunteers to inform sample population characteristics.
Concussion history data | Baseline
  Participant concussion history will provide descriptive analysis of mechanism of injury, number of concussions, characteristics of current concussion injury (time since injury, hospitalization due to injury)

CONTACTS AND LOCATIONS:
Overall Officials: James P Dickey, PhD, Principal Investigator — Western University
Locations (1):
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Each participant will be identified with a code based on study protocol, testing year and participant number (e.g., SP#YYPID#: SP#201001) that correlates to his or her addition to the study. The master reference that contains the decoding system will be stored on a secure server behind fire wall protection. All other data will be labeled using the participant's identification code.

REFERENCES:
- [Background] Milosevic I, Levy HC, Alcolado GM, Radomsky AS. The Treatment Acceptability/Adherence Scale: Moving Beyond the Assessment of Treatment Effectiveness. Cogn Behav Ther. 2015;44(6):456-69. doi: 10.1080/16506073.2015.1053407. Epub 2015 Jun 19. PMID 26091250
- [Background] Eyres S, Carey A, Gilworth G, Neumann V, Tennant A. Construct validity and reliability of the Rivermead Post-Concussion Symptoms Questionnaire. Clin Rehabil. 2005 Dec;19(8):878-87. doi: 10.1191/0269215505cr905oa. PMID 16323387
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171